CLINICAL TRIAL: NCT07000162
Title: LAttice Radiation Therapy for Large Lesions: Reggio Emilia Single-arm Phase II Trial (LART Trial)
Brief Title: LAttice Radiation Therapy for Large Lesions: Reggio Emilia Single-arm Phase II Trial
Acronym: LART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5/2025/SPER/IRCCSRE
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Palliative Radiotherapy
Keywords: Lattice radiotherapy; Lattice radiation therapy; Spatially Fractionated Radiation Therapy; Large cancers; Palliative radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lattice radiation therapy (Experimental): Radiation: A total dose will be 20 Gy, with a simultaneous boost to selected tumor regions (hot spots) reaching a minimum median dose of 50 Gy.
  Interventions: Radiation: Lattice radiation therapy

INTERVENTIONS:
Radiation: Lattice radiation therapy — A total dose will be 20 Gy, with a simultaneous boost to selected tumor regions (hot spots) reaching a minimum median dose of 50 Gy.
  Peripheral blood (PB) samples for the immune cell characterization and quantification of immune-related circulating factors will be collected at baseline (pre-therapy) and within 7 -14 days after the end of the treatment (post-therapy).

SUMMARY:
This study evaluates the activity and toxicity of Lattice Radiation Therapy (LRT) in patients with large, unresectable non-brain neoplastic lesions requiring palliative treatment. Eligible patients will 5 fractions LRT, delivered in every other day, to 20 Gy with a simultaneous boost to a minimum median dose of 50 Gy. No concomitant antineoplastic drugs will be allowed. Patients will be followed at 14, 30, 60, and 90 days after treatment, then every 3 months up to 1 year. Tumor response will be assessed using objective response rate (ORR) per RECIST 1.1, with CT scans at 3, 6, 9, and 12 months. Secondary endpoints include local control, toxicity (CTCAE v.5.0), and patient-reported outcomes (PROMs) to assess their quality of life (EORTC QLQ-C15-PAL and PRO-CTCAE). Exploratory objectives will assess the immunomodulatory effects of LRT through immune cell characterization and quantification of immune-related circulating factors before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 on day signing informed consent
* Histologically or cytologically confirmed cancer.
* Performance status of 0-2 on the ECOG Performance Scale.
* Advanced or locally advanced disease, not eligible for curative-intent treatment.
* Life expectancy > 6 months.
* At least one measurable non-brain site of disease with a diameter ≥ 4.5 cm, in any direction
* Ability to understand and willingness to sign the written informed consent document (or that of legally authorized representative, if applicable).

Reproductive Status

* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of LRT.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of LRT plus 30 days (duration of ovulatory cycle).
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of LRT plus 90 days (duration of sperm turnover).
* Investigators shall counsel WOCBP patients and male patients who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy

Exclusion Criteria:

* Additional malignancy that is progressing or requires active treatment. Exceptions include basal and squamous cell carcinoma of the skin or in situ cervical
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of the start of LRT.
* Prior high-dose radiotherapy overlapping with any planned site of protocol radiotherapy, if the dose overlap is > 10 Gy or is determined not safe by the treating physician.
* HIV patients with CD4+ T-cell counts < 350 cells/mcL or with a history of AIDS-defining opportunistic infection, within the 12 months prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | At 3 months following completion of Lattice radiation therapy
  Percentage of patients with complete and partial response according to RECIST1.1 criteria

SECONDARY OUTCOMES:
Local Control | At 3, 6,9, and 12 months following completion of Lattice radiation therapy.
  Percentage of patients with complete response, partial response, and stable disease according to RECIST1.1 criteria
Treatment-related toxicity | 1 year following completion of Lattice radiation therapy.
  Percentage of patients with treatment-related adverse events measured by CTCAE version 5.0
Patient-reported outcomes (Quality of life) | 2 weeks, 30 days, 60 days, and 90 days, 6 months, 9 months, 1 year
  Scores modification compared to baseline at questionnaire EORTC QLQ-C15-PAL (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 15 - Palliative care version), a 15-item scale with scores ranging from 0 to 100. Higher scores on functional and global health status scales indicate better quality of life, while higher scores on symptom scales indicate worse symptom burden.
Patient-reported outcomes (Quality of life) | 2 weeks, 30 days, 60 days, and 90 days, 6 months, 9 months, 1 year
  Scores modification compared to baseline at questionnaire PRO-CTCAE (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events), a patient-reported outcome measure developed by the U.S. National Cancer Institute. Each item is scored on a 5-point scale (range: 0-4), where higher scores indicate greater symptom frequency, severity, or interference with daily activities.

OTHER OUTCOMES:
Immunomodulatory effects of Lattice Radiation Therapy (LRT) | 7-14 days after the end of the treatment
  Modification compared to baseline of immune cells through cell immunophenotyping and immune-related circulating factors possibly associated with LRT compared to baseline (Exploratory Outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Iotti, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan W, Khan MK, Wu X, Simone CB 2nd, Fan J, Gressen E, Zhang X, Limoli CL, Bahig H, Tubin S, Mourad WF. Spatially fractionated radiation therapy: History, present and the future. Clin Transl Radiat Oncol. 2019 Oct 22;20:30-38. doi: 10.1016/j.ctro.2019.10.004. eCollection 2020 Jan. No abstract available. PMID 31768424
- [Background] Wu X, Perez NC, Zheng Y, Li X, Jiang L, Amendola BE, Xu B, Mayr NA, Lu JJ, Hatoum GF, Zhang H, Chang SX, Griffin RJ, Guha C. The Technical and Clinical Implementation of LATTICE Radiation Therapy (LRT). Radiat Res. 2020 Dec 1;194(6):737-746. doi: 10.1667/RADE-20-00066.1. PMID 33064814
- [Background] Duriseti S, Kavanaugh J, Goddu S, Price A, Knutson N, Reynoso F, Michalski J, Mutic S, Robinson C, Spraker MB. Spatially fractionated stereotactic body radiation therapy (Lattice) for large tumors. Adv Radiat Oncol. 2021 Jan 8;6(3):100639. doi: 10.1016/j.adro.2020.100639. eCollection 2021 May-Jun. PMID 34195486
- [Background] Iori F, Cappelli A, D'Angelo E, Cozzi S, Ghersi SF, De Felice F, Ciammella P, Bruni A, Iotti C. Lattice Radiation Therapy in clinical practice: A systematic review. Clin Transl Radiat Oncol. 2022 Dec 20;39:100569. doi: 10.1016/j.ctro.2022.100569. eCollection 2023 Mar. PMID 36590825
- [Background] Duriseti S, Kavanaugh JA, Szymanski J, Huang Y, Basarabescu F, Chaudhuri A, Henke L, Samson P, Lin A, Robinson C, Spraker MB. LITE SABR M1: A phase I trial of Lattice stereotactic body radiotherapy for large tumors. Radiother Oncol. 2022 Feb;167:317-322. doi: 10.1016/j.radonc.2021.11.023. Epub 2021 Dec 4. PMID 34875286
- [Background] Asur R, Butterworth KT, Penagaricano JA, Prise KM, Griffin RJ. High dose bystander effects in spatially fractionated radiation therapy. Cancer Lett. 2015 Jan 1;356(1):52-7. doi: 10.1016/j.canlet.2013.10.032. Epub 2013 Nov 15. PMID 24246848
- [Background] Kumari S, Mukherjee S, Sinha D, Abdisalaam S, Krishnan S, Asaithamby A. Immunomodulatory Effects of Radiotherapy. Int J Mol Sci. 2020 Oct 31;21(21):8151. doi: 10.3390/ijms21218151. PMID 33142765
- [Background] Kanagavelu S, Gupta S, Wu X, Philip S, Wattenberg MM, Hodge JW, Couto MD, Chung KD, Ahmed MM. In vivo effects of lattice radiation therapy on local and distant lung cancer: potential role of immunomodulation. Radiat Res. 2014 Aug;182(2):149-62. doi: 10.1667/RR3819.1. Epub 2014 Jul 18. PMID 25036982
- [Background] Ferini G, Valenti V, Tripoli A, Illari SI, Molino L, Parisi S, Cacciola A, Lillo S, Giuffrida D, Pergolizzi S. Lattice or Oxygen-Guided Radiotherapy: What If They Converge? Possible Future Directions in the Era of Immunotherapy. Cancers (Basel). 2021 Jun 30;13(13):3290. doi: 10.3390/cancers13133290. PMID 34209192